CLINICAL TRIAL: NCT00803504
Title: Correlation of Optic Disk Morphology and Ocular Perfusion Parameters in Patients With Primary Open Angle Glaucoma
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Other Study IDs: OPHT-120905
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Primary Open Angle Glaucoma
Keywords: optic disc morphology; ocular blood flow; retina; ocular physiology
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: ocular blood flow measurement

SUMMARY:
Glaucoma is one of the most common causes of blindness in the industrialized nations. For a long time glaucoma has been defined as a disease in which high intraocular pressure (IOP) leads to irreversible optic disc damage and subsequent visual field loss. However, recent investigations show that IOP is not the only factor that is involved in the glaucomatous process leading to retinal ganglion cell death. The role of vascular factors in the pathogenesis of glaucoma has recently received much attention based on animal experiments and epidemiological studies. It is, however, assumed that vascular factors do not contribute to same degree in all glaucoma patients. Generally, it is believed that a vascular component is more important in normal tension glaucoma patients and patients with underlying cardiovascular disease. Little is, however, known about a potential association between optic nerve head morphology and ocular perfusion in POAG patients. The current study seeks to gain insight into this association by assessing ocular blood flow parameters with a number of noninvasive technologies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years
* Unilateral or bilateral primary open angle glaucoma
* At least 3 reliable visual field tests showing CPSD >= 2.0 in the eye that will be studied

Exclusion Criteria:

* History of acute angle closure
* Closed or barely open anterior chamber angle
* Standard deviation of visual field testing > 10
* Intraocular surgery or argon laser trabeculoplasty within the last six months
* Ocular inflammation or infection within the last three months
* Topical or systemically/oral therapy with steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow (scanning laser Doppler flowmetry, laser Doppler flowmetry)
Retinal blood flow (scanning laser Doppler flowmetry, laser Doppler velocimetry + retinal vessel analyzer)
Choroidal blood flow (laser Doppler flowmetry, laser interferometry, pneumotonometry)
Optic nerve head morphology parameters
Fundus photography: evaluation based on Jonas et al. 2003 J Glaucoma 12:260-265,
Heidelberg Retina Tomograph: evaluation based on Iester et al. 2001 Am J Ophthalmol 132: 57-62,

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Deparmtent of Clinical Pharmacology, Vienna, Austria